CLINICAL TRIAL: NCT02134665
Title: Unexpected Pharmacokinetics of Vancomycin in Patients With Severe Acute Pancreatitis Compared With Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, He Juan, Miss, Ruijin Hospital
Other Study IDs: hejuanwin19811119
Record Dates: First submitted 2014-01-24; First posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Arbitrary Restriction Polymorphism 1
Keywords: Vancomycin; severe acute pancreatitis; Creatinine clearance
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- severe acute pancreatitis: patients who received vancomycin therapy and whose serum vancomycin level was monitored, and who also had diagnosed as severe acute pancreatitis.
- Pneumonia: patients who received vancomycin therapy and whose serum vancomycin level was monitored, and who also had diagnosed as pneumonia.

SUMMARY:
The purpose of this study was to evaluate the influence of severe acute pancreatitis on the serum level of vancomycin, a glycopeptide antibacterial agent.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the influence of severe acute pancreatitis on the serum level of vancomycin, a glycopeptide antibacterial agent.

After reviewing more than 6000 clinical charts of patients who received vancomycin therapy and whose serum vancomycin level was monitored between January 2010 and December 2013, we identified 212 patients who also had diagnosed as severe acute pancreatitis (SAP group), and 98 patients who also had diagnosed as pneumonia (pneumonia group) at that time. The fluorescence polarization immunoassay method was used to measure vancomycin serum trough concentrations in these patients 30 min before the next administration. Using these measurements, we calculated the pharmacokinetic parameters using the Bayesian estimator.

ELIGIBILITY:
Inclusion Criteria:

* age 18-85years old
* vancomycin use ≥ 3days

Exclusion Criteria:

* age <18years old or >85 years old
* vancomycin use < 3days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who used vancomycin and who had diagnosed as severe acute pancreatitis (SAP group), and patients who had diagnosed as pneumonia (pneumonia group) . meanwhile, the fluorescence polarization immunoassay method was used to measure vancomycin serum trough concentrations in these patients 30 min before the next administration.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
vancomycin serum trough concentrations in these patients just prior to the next vancomycin serum trough concentrations was measured | patients will be followed for the duration of hospital stay, an expected average of 5 weeks
  vancomycin serum trough concentrations was measured in patients just prior to the next dose at steady-state conditions (approximately after the fourth dose).

SECONDARY OUTCOMES:
the pharmacokinetic parameters was calculated using the Bayesian estimator. | patients will be followed for the duration of hospital stay, an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Hua Yang, Prof., Study Director — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China